CLINICAL TRIAL: NCT04319510
Title: Supportive Effects of Craniosacral Therapy for Women With Breast Cancer: a Randomized Controlled Trial
Brief Title: Supportive Effects of Craniosacral Therapy for Women With Breast Cancer
Acronym: CRANIO4US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Heidemarie Haller, Principal Investigator, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2019402
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Complementary Therapies
Keywords: Craniosacral Therapy; Breast cancer; Randomized Controlled Trial; Self-help strategies; Self-efficacy; Coping
MeSH Terms: conditions — Breast Neoplasms | interventions — Therapeutics; Waiting Lists

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator who will perform the group assignment will have no contact to the study participants. The outcome assessors will be blinded to group allocation. The statistician who will perform the analyses will kept blind to the group intervention by renaming groups with numbers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Craniosacral therapy (Experimental): 24 CST units à 45 minutes over 12 weeks. Follow-up assessment 6 months after randomization.
  Interventions: Procedure: Craniosacral therapy
- Craniosacral self-help group training (Experimental): 24 CST units à 45 minutes over 12 weeks. Follow-up assessment 6 months after randomization.
  Interventions: Procedure: Craniosacral self-help group training
- Treatment as usual / wait list control (Other): Waiting period of six months.
  Interventions: Procedure: Treatment as usal / wait list

INTERVENTIONS:
Procedure: Craniosacral therapy — The first experimental group of patients will receive 24 units à 45 minutes over 12 weeks (2 consecutive units per week) offered by a trained craniosacral therapist within a 1:1 setting. Treatment as usual is allowed.
  Arms: Craniosacral therapy
Procedure: Craniosacral self-help group training — The second experimental group of patients will receive 24 teaching units (TUs) à 45 minutes over 12 weeks offered by a trained craniosacral therapist within a group setting. The group training will start with an introductory day (8 TUs), followed by 6 practice evenings every two weeks (2 TUs each) and a final afternoon (4 TUs). The patients have to agree to participate in the introductory day and 90% of the following TUs. All patients will receive a script with theoretical CST information and descriptions of the learned techniques, which should facilitate the correct practice at home. Treatment as usual is allowed.
  Arms: Craniosacral self-help group training
Procedure: Treatment as usal / wait list — The control group will receive no specific study treatment for a waiting period of six months. Treatment as usual is allowed. Afterwards they were offered self-selection to 1:1 CST or participation in the CST self-help group training.
  Arms: Treatment as usual / wait list control

SUMMARY:
Craniosacral Therapy (CST) is a non-manipulative, very gentle, manual treatment method that aims to release restrictions of the fasciae and regulate the arousal of the sympathetic nervous system, which is often increased in chronically ill patients. Initial randomized trials support CST's efficacy and effectiveness in reducing symptoms of patients with psychosomatic and chronic pain disorders. To date, there is no trial investigating the effectiveness of CST as a supportive strategy for enhancing cancer-related quality of life in women with breast cancer. In clinical practice, therapists also report alleviating as well as regulating effects of simple CST self-help techniques, offered to patients within a group concept.

Within the recent study, a CST treatment and self-help protocol for women after curative therapy of breast cancer was developed and shall be tested against a waiting list control group. The first group will receive 24 units of CST treatment in a 1:1 setting with a certified craniosacral therapist over 12 weeks. The second group will receive 24 units of group training in CST self-help techniques offered by a certified craniosacral therapist over 12 weeks. They will be reassessed after 12 and 26 weeks (6 months) after randomization. The third group will wait for 26 weeks and will receive no specific study intervention. After 26 weeks patients of the third group were offered self-selection to either individual CST or CST self-help group training. For all groups, treatment as usual is allowed.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer (stage I-III) survivors after finishing curative chemotherapy and/or radiation
* Impaired breast caner-related quality of life (< 112,8 points on the FACT-B)

Exclusion Criteria:

* Planned surgery, adjuvant therapy (chemotherapy and/or radtiation), or rehabilitation during the study period
* Pregnancy
* Simultaneous participation in other clinical trials

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Breast cancer-related quality of life - total score | week 12
  Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) Questionnaire: The FACT-B consists of 37 self-report items and assesses the specific breast cancer-related quality of life as a total score of 4 general and 1 breast-cancer specific subscale. A higher score indicates a higher cancer-related quality of life.

SECONDARY OUTCOMES:
Breast cancer-related quality of life - sub scores | week 12
  Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) Questionnaire: The FACT-B consists of 37 self-report items and assesses the specific breast cancer-related quality of life on 4 general and 1 breast-cancer specific subscale. A higher score indicates a higher cancer-related quality of life.
Breast cancer-related quality of life - total score | week 26
  Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) Questionnaire: The FACT-B consists of 37 self-report items (4 general subscales and one breast-cancer specific subscale, which will be summarized to a total score) and assesses the specific breast cancer-related quality of life. A higher score indicates a higher cancer-related quality of life.
Breast cancer-related quality of life - sub scores | week 26
  Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) Questionnaire: The FACT-B consists of 37 self-report items and assesses the specific breast cancer-related quality of life on 4 general and 1 breast-cancer specific subscale. A higher score indicates a higher cancer-related quality of life.
Fatigue | week 12
  Functional Assessment of Cancer Therapy - Fatigue (FACT-F) Questionnaire: The addoitional F-scale of the FACT consists of 13 self-report items and assesses fatigue related to cancer on 1 scale. A higher score indicates a higher cancer-related fatigue.
Fatigue | week 26
  Functional Assessment of Cancer Therapy - Fatigue (FACT-F) Questionnaire: The addoitional F-scale of the FACT consists of 13 self-report items and assesses fatigue related to cancer on 1 scale. A higher score indicates a higher cancer-related fatigue.
Endocrine symptoms | week 12
  Funcitonal Assessment of Cancer - Endocrine Symptom (FACT-ES) Questionnaire: The additonal ES-scale of the FACT consists of 19 self-report items and assesses symptoms related to the endocrine system / antihormonal therapy on 1 scale. A higher score indicates a higher endocrine symptoms.
Endocrine symptoms | week 26
  Funcitonal Assessment of Cancer - Endocrine Symptom (FACT-ES) Questionnaire: The additonal ES-scale of the FACT consists of 19 self-report items and assesses symptoms related to the endocrine system / antihormonal therapy on 1 scale. A higher score indicates a higher endocrine symptoms.
Sleep disturbance | week 12
  Patient related outcomes measurement information system - sleep disturbance (PROMIS-SD) Short form: The SD-short form of the PROMIS consists of 8 self-report items and assesses the disturbance of sleep on 1 scale. A higher score indicates higher disturbances of the sleep.
Sleep disturbance | week 26
  Patient related outcomes measurement information system - sleep disturbance (PROMIS-SD) Short form: The SD-short form of the PROMIS consists of 8 self-report items and assesses the disturbance of sleep on 1 scale. A higher score indicates higher disturbances of the sleep.
Severity of insomnia | week 12
  Insomnia Severity Index (ISI): The ISI consists of 7 self-report items and assesses the severity of insomnia on 1 scale. A higher score indicates higher severity of insomnia.
Severity of insomnia | week 26
  Insomnia Severity Index (ISI): The ISI consists of 7 self-report items and assesses the severity of insomnia on 1 scale. A higher score indicates higher severity of insomnia.
State anxiety | week 12
  Patient related outcomes measurement information system - anxiety/emotional distress (PROMIS-A/ED) Short form: The A/ED-short form of the PROMIS consists of 7 self-report items and assesses state anxiety on one scale. A higher score indicates higher anxiety.
State anxiety | week 26
  Patient related outcomes measurement information system - anxiety/emotional distress (PROMIS-A/ED) Short form: The A/ED-short form of the PROMIS consists of 7 self-report items and assesses state anxiety on one scale. A higher score indicates higher anxiety.
Fear of recurrence | week 12
  The Fear of Relapse/Recurrence Scale (FRRS): The FRRS consists of 5 self-report items and assesses the fear of cancer recurrence on one scale. A higher score indicates higher fear of recurrence.
Fear of recurrence | week 26
  The Fear of Relapse/Recurrence Scale (FRRS): The FRRS consists of 5 self-report items and assesses the fear of cancer recurrence on one scale. A higher score indicates higher fear of recurrence.
Severity of depressive symptoms | week 12
  Center for epdiemiologic studies depression scale (CES-D): The CES-D consists of 10 self-report items and assesses the severity of depressive symptoms on one scale. A higher score indicates higher severity of depressive symptoms.
Severity of depressive symptoms | week 26
  Center for epdiemiologic studies depression scale (CES-D): The CES-D consists of 10 self-report items and assesses the severity of depressive symptoms on one scale. A higher score indicates higher severity of depressive symptoms.
Number of patients with adverse events | week 12
  The number of patients with adverse events and serious adverse events will be recorded according to the Common Terminology Criteria for Adverse Events (CTCAE)
Number of patients with adverse events | week 26
  The number of patients with adverse events and serious adverse events will be recorded according to the Common Terminology Criteria for Adverse Events (CTCAE)
Total number, type, and grade of adverse events | week 12
  The total number, type and grade of adverse events and serious adverse events will be recorded according to the Common Terminology Criteria for Adverse Events (CTCAE)
Total number, type, and grade of adverse events | week 26
  The total number, type and grade of adverse events and serious adverse events will be recorded according to the Common Terminology Criteria for Adverse Events (CTCAE)

OTHER OUTCOMES:
Expectations about treatment efficacy | week 0
  Treatment Credibility Scale (TCS): The TCS consists of 4 self-report items, which are answered on a Numeric Rating Scale (NRS). One item asks about the expectations of efficacy of the study treatments and 3 items about treatment credibility (see below). A higher score indicates higher treatment expectations.
Expectations about self-efficacy | week 0
  Numeric Rating Scale (NRS): Expectations about the self-efficacy of performing the learned CST techniques at home were assessed using a self-report NRS. A higher score indicates higher expectations of self-efficacy.
Treatment Credibility | week 12
  Treatment Credibility Scale (TCS): The TCS consists of 4 self-report items, which are answered on a Numeric Rating Scale (NRS). One item asks about the expectations of efficacy of the study treatments (se above) and 3 items about treatment credibility. A higher score indicates higher treatment credibility.
Relation between therapist and patient | week 12
  Helping Alliance Questionnaire (HAQ): The HAQ consists of 11self-report items and assesses the therapeutic relation on two subscales: quality of the therapeutic relation and satisfaction with the treatment. A higher score indicates a higher quality of the therapeutic relation / a higher satisfaction with the treatment.
Actually received social support | week 12
  Berlin Social Support Scales - Actually Received Support (BSSS-ARS) subscale: The BSSS-ARS consists of 15 self-report items and assesses the actually received social support on 4 subscales: emotional support, instrumental support, informational support, and satisfaction with support. A higher score indicates higher received social support.
Actually received social support | week 26
  Berlin Social Support Scales - Actually Received Support (BSSS-ARS) subscale: The BSSS-ARS consists of 15 self-report items and assesses the actually received social support on 4 subscales: emotional support, instrumental support, informational support, and satisfaction with support. A higher score indicates higher received social support.
Body Awareness | week 12
  Body Responsiveness Questionnaire (BRQ): The BRQ consists of 7 self-report items and assesses body awareness on 3 subscales: Importance of Interoceptive Awareness, Perceived Connection, and Suppression of Bodily Sensations. A higher score indicates higher body awareness on the subscales Importance of Interoceptive Awareness and Perceived Connection, while a higher score indicates lower body awareness on the subscale Suppression of Bodily Sensations.
Body Awareness | week 26
  Body Responsiveness Questionnaire (BRQ): The BRQ consists of 7 self-report items and assesses body awareness on 3 subscales: Importance of Interoceptive Awareness, Perceived Connection, and Suppression of Bodily Sensations. A higher score indicates higher body awareness on the subscales Importance of Interoceptive Awareness and Perceived Connection, while a higher score indicates lower body awareness on the subscale Suppression of Bodily Sensations.
Interview | week 12
  Semi-structured interview: A pre-developed semi-structured interview guide asks about the personal experiences with the effects and safety of craniosacral therapy/self-help techniques.
Craniosacral-specific quality of life | week 12
  Warwick Holistic Health Questionnaire (WHHQ): The WHHQ consists of 25 self-report items and assesses craniosacral-specific quality of life on one scale. A higher score indicates higher craniosacral-specific quality of life. The German version of the WHHQ shall be validated within this trial.
Craniosacral-specific quality of life | week 26
  Warwick Holistic Health Questionnaire (WHHQ): The WHHQ consists of 25 self-report items and assesses craniosacral-specific quality of life on one scale. A higher score indicates higher craniosacral-specific quality of life. The German version of the WHHQ shall be validated within this trial.
Duration of homework | week 1-12
  The duration of performing the CST techniques at home (for group 2) will be assessed using a diary.

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, Prof. MD, Study Director — Center for Integrative Medicine and Planetary Health, University Hospital Essen, University of Duisburg-Essen
Locations (3):
- Germany (3):
  - Center for Integrative Medicine and Planetary Health, University Hospital Essen, University of Duisburg-Essen, Essen
  - Breast Unit, Evang. Kliniken Essen-Mitte, Essen
  - Department of Gynecology and Obstetrics, University Hospital Essen, University of Duisburg-Essen, Essen

IPD SHARING:
Plan to Share IPD: No